CLINICAL TRIAL: NCT06282718
Title: Perpetual Observational Study (POS) of Acute Respiratory Infections (ARI) in Primary Care Settings (PC) Across Europe
Brief Title: A Long-term Observational Study Evaluating the Presentation and Management of Acute Respiratory Tract Infections in Primary Care Across Europe
Acronym: POS-ARI-PC
Status: Recruiting | Type: Observational
Sponsor: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Collaborators: UMC Utrecht (Other); University of Oxford (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: POS-ARI-PC CORE and AUDIT; 965313 (Other Grant/Funding Number: European Union); 10204126 (Registry Identifier: ISRCTN); 55487 (Other: NIHR CPMS); 324504 (Other: IRAS)
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Acute Respiratory Tract Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A combined throat/nose swab sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- POS-ARI-PC: POS-ARI-PC AUDIT:
  Anonymous registration of patients of any age presenting at the participating primary care facility with ARI.
  POS-ARI-PC CORE:
  Patients of any age presenting at the participating primary care facility with ARI.
  POS-ARI-PC-001:
  Patients 60 and over, or aged 50 to 59 years and have a long-term health condition which makes them eligible for the yearly influenza vaccination under the national influenza vaccination programme, presenting at the participating primary care facility with ARI.

SUMMARY:
Acute respiratory infection (ARI) is the commonest reason for consulting in community care. Furthermore, new and re-emerging pathogens are often first noticed in primary care (PC). The POS-ARI-PC study is a long-term study, with the aim of describing the nature of ARI in adults and children presenting to PC across Europe. The POS-ARI-PC study will provide critically important data on the presentation and management of ARI, and build a research-ready infrastructure for studies related to the treatment, diagnosis, and prevention of ARI in primary care settings. Additional observational studies will be embedded and use the infrastructure developed in POS-ARI-PC.

DETAILED DESCRIPTION:
The main aim for POS-ARI-PC is to provide a platform for continuous data capture for patients with ARI presenting to primary care settings across Europe, covering cases caused by known and emerging respiratory pathogens with epidemic and pandemic potential, in order to generate observational evidence to inform care and maintain study- readiness for RCT evaluations. The POS-ARI-PC platform will thereby support the efficient set-up of new clinical studies and trials, which will be embedded into the platform.

We have developed two overarching protocols for the POS-ARI-PC. The POS-ARI-PC AUDIT protocol allows for a flexible annual anonymous prospective audit-type registration to describe the presentation and management of patients presenting in primary care with ARI. This provides the infrastructure for patient sampling and follow-up, and in which randomisation can be activated for platform trials to evaluate a range of interventions that can be added and replaced over time. This has resulted in the POS-ARI-PC CORE protocol.

POS-ARI-PC AUDIT:

This is a flexible annual anonymous prospective audit-type registration to describe the presentation and management of patients presenting in primary care with ARI. POS-ARI-PC AUDIT will be delivered through a prospective, multi-country, audit-type anonymous registration of presentation and management of approximately 2,000 patients presenting to PC annually across Europe. This audit will benchmark the case mix and care of patients consulting in PC. These can include general practice, urgent care centres, accident and emergency and other acute services in hospitals, for adult and paediatric patients, both in and out of office hours.

POS-ARI-PC CORE:

This is a non-randomised, prospective, observational study of the presentation, management, microbiology and outcome of acute respiratory tract infection in primary care.

POS-ARI-PC CORE has the following three objectives:

Objective 1. A prospective, observational study of ARI patients in primary care to undergo study-specific sampling upon inclusion and be followed up for 28 days to capture the aetiology of their ARI and describe clinical outcomes.

Objective 2. A qualitative study with research professionals, clinicians, and patients to a) gain a deep understanding of the research process, and the meaning of results and to identify barriers and opportunities for implementation of changes considering findings, and b) explore the views and experiences of patients who consult European primary care services for ARI symptoms since the COVID-19 pandemic.

Objectives 3. To ensure research readiness for including embedded observational and randomised evaluations to answer questions about the effectiveness of diagnostic, behavioural or therapeutic management strategies for ARI in PC. When a new embedded observational study or RCT is added to the POS-ARI-PC a study-specific appendix (SSA) or an intervention-specific appendix (ISA) will be developed which details the (changes in) the study population, the research question, objectives, outcomes, study-specific processes and analysis. This will be appended to the POS-ARI-PC CORE Protocol and all appropriate approvals will be gained for each SSA or ISA.

Participation in the study will last for 28 days. Once consented to the study, a member of the study team will complete a short questionnaire collecting the participants' names and contact information, some details about them, and the symptoms they have been experiencing. A combined throat/nose swab will be collected from the patient for study purposes.

Participants will also be asked to tell us about how they are feeling today and for the next 14 days via an online or paper daily diary. They might be telephoned to ask some questions if they are unable to complete the daily diary. Their GP will be contacted after day 28 to collect information about their consultations and hospital referrals in the 28-day period.

A small number of enrolled participants who consented (optional) to be contacted by the research team about the nested qualitative study will be invited for a process evaluation interview.

POS-ARI-PC-001:

The first embedded study, POS-ARI-PC-001, will be conducted as a prospective observational study to estimate the incidence of medically-attended RSV, HMPV, HPIV and RV infections in an elderly population. This embedded study is appended to the POS-ARI-PC CORE Protocol as a study specific appendix (SSA).

ELIGIBILITY:
POS-ARI-PC AUDIT:

Inclusion Criteria:

Eligible patients will be of any age consulting (telephone, video, face-to-face) with a participating health care facility with:

* Symptoms suggestive of an acute lower RTI with cough as predominant symptom and with illness duration less than 28 days, AND/OR
* Symptoms suggestive of an acute upper RTI with sore throat and/or coryza as predominant symptom and with illness duration of less than 14 days AND/OR
* Patients otherwise suspected of COVID-19, influenza or RSV.

Exclusion Criteria:

Patients will not be eligible for if they have withdrawn their consent for anonymous data collection for research by their health care facility.

POS-ARI-PC CORE:

Inclusion criteria:

Eligible patients will be of any age consulting (telephone, video, face to face) with a participating primary health care facility with:

* Symptoms suggestive of an acute lower respiratory infection with cough as the predominant symptom, with illness duration less than 28 days, AND/OR
* Symptoms suggestive of an acute upper respiratory infection with sore throat and/or coryza as the predominant symptom, with illness duration of less than 14 days AND/OR
* Other symptoms suggestive of COVID-19, Influenza, RSV AND
* Participant or legal guardian(s) willing and able to provide informed consent and comply with study procedures

Exclusion criteria:

Patients will not be eligible if:

* According to the judgement of the recruiting clinician, they will not be able comply with study procedures, for example because they do not understand the language in which the study is being conducted locally (and have no one to help and translate for them); have a serious psychiatric disorder; or are terminally ill
* Symptoms of presumed non-infective origin
* Participant requires admission to hospital on the day of inclusion

Additional in/exclusion criteria might apply to embedded studies and will be described in the SSA or ISA.

POS-ARI-PC-001:

Symptoms and Duration Symptoms suggestive of an acute lower RTI with new or increased cough as the predominant symptom, with illness duration ≤10 days; AND/OR Symptoms suggestive of an acute upper RTI with sore throat and/or coryza as the predominant symptom, with illness duration ≤10 days;

Age Aged 60 years and over OR Aged 50 to 59 years and have a long-term health condition which makes them eligible for the yearly influenza vaccination under the national influenza vaccination programme;

Consent Willing and able to provide informed consent and have a swab taken.

Exclusion Criteria:

As per the POS-ARI-PC CORE Protocol, with one exception: patients needing hospitalisation can be recruited into the study if timing allows. Patients can provide a swab and decide not to participate in the follow-up procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age group presenting to primary care settings with an ARI.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Age Bands | Baseline (Day 0)
  Participant age recorded at baseline by site study team.
The proportion with a preliminary diagnosis of various sub-categories of ARI (e.g. LRTI, URTI) | Baseline (Day 0)
  Working diagnosis recorded at baseline by site study team.
Overall illness severity rating | Baseline (Day 0)
  Overall illness severity (clinician's impression) recorded at baseline (mild, moderate or severe) by site study team.
Swab samples taken and retrospective viral/microbiological infection analysis performed (multiplex PCR) to identify potential causative pathogens. | Baseline (Day 0)
  Participants have a combined oropharyngeal and nasal swab taken at the baseline visit which will be subjected to PCR-based analysis to identify potential causative pathogens.
Proportion undergoing POC (with results) and lab-based investigations | Baseline (Day 0) and day 28.
  POC investigations recorded at baseline and results recorded at day 28 by site study team.
Details of prescriptions given on presentation of ARI | Baseline (Day 0)
  Prescriptions given at presentation recorded at Baseline by site study team.
Details of tests ordered on presentation of ARI | Baseline (Day 0)
  Tests ordered at presentation recorded at Baseline by site study team.
Return to usual daily activities | Day 1-14
  Participants asked if they have returned to usual activities in daily diary.
Feeling recovered from RTI | Day 1-14
  Participants asked if they are feeling recovered from RTI in daily diary.
Use of prescription medication | Day 1-14
  Participants asked if they have used prescription medication for the RTI in daily diary.
Use of over the counter medications | Day 1-14
  Participants asked if they have used over the counter medication for the RTI in daily diary.
Complications reported associated to ARI presentation | Day 28
  Recorded at day 28 by a member of the site study team.
Variation in practice and advice from national guidelines, to be fed back to national teams | Baseline (Day 0)
  Practice and advise recorded at Baseline by site study team.

SECONDARY OUTCOMES:
Recommendations on how to improve study processes, recruitment and study communication based on shared understanding and insights from researchers, clinicians, and patients. | After day 28
  Using qualitative research methods, interviews conducted with research professionals, clinicians and patients to gain a deep understanding of the research process, meaning of results and to identify barriers and opportunities for implementation of findings. Capturing patients' views on their vulnerability towards ARI in the community since the COVID19 pandemic.
An understanding of the meaning of study results for European primary care, from the perspectives of clinicians and patients, and recommendations regarding the implementation of findings. | After day 28
  Using qualitative research methods, interviews conducted with research professionals, clinicians and patients to gain a deep understanding of the research process, meaning of results and to identify barriers and opportunities for implementation of findings. Capturing patients' views on their vulnerability towards ARI in the community since the COVID19 pandemic.
An understanding of changing health-seeking behaviour, management and expectations to inform clinical studies and trials | After day 28
  Measured using an interview conducted by the social science team after taking part in the main study and using a descriptive analysis
Approval for a study-specific appendix (SSA) or an intervention-specific appendix (ISA) of an embedded (non) randomised study for ARI in primary care associated with this POS, measured using the number of embedded studies to this POS-ARI-PC platform over | Through study completion
  To ensure research readiness for including embedded observational and randomised evaluations to answer questions about the effectiveness of diagnostic, behavioural or therapeutic management strategies for ARI in PC.

CONTACTS AND LOCATIONS:
Locations (3):
- Universiteit Antwerpen, Antwerp, Belgium
- Centre Hospitalier Universitaire de Limoges, Limoges, France
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No